CLINICAL TRIAL: NCT07161895
Title: Prevalence of Kinesiophobia and Its Effects on Functional Capacity and Pain Severity in Patients With Primary Knee Osteoarthritis
Brief Title: Kinesiophobia and Its Impact on Pain and Function in Knee Osteoarthritis
Acronym: KinesiOA
Status: Completed | Type: Observational
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nadide Koca, Principal Investigator, Ankara Training and Research Hospital
Other Study IDs: AnkaraTRH-FTR-NK-08; E-25-543 (Other: Ankara Training and Research Hospital Ethics Committee)
Record Dates: First submitted 2025-08-31; First posted 2025-09-09 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis (Knee OA); OA; Kinesiophobia
Keywords: Kinesiophobia; Pain; Functional Capacity; WOMAC; Visual Analogue Scale (VAS); Tampa Scale for Kinesiophobia (TSK); Kellgren-Lawrence Grading
MeSH Terms: conditions — Osteoarthritis, Knee; Kinesiophobia; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Knee Osteoarthritis Patients: Adults aged 40-85 years with radiographically confirmed primary knee osteoarthritis. Participants will complete clinical examination, Kellgren-Lawrence radiographic grading, Visual Analogue Scale (VAS) for pain, Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) for function, and Tampa Scale for Kinesiophobia (TSK). Assessments are performed at a single visit; no interventions are applied.

SUMMARY:
Knee osteoarthritis (OA) is the most common chronic joint disorder, especially in older adults, and is a leading cause of pain, disability, and reduced quality of life. Patients with OA often experience pain and functional limitations that may contribute to psychological factors such as anxiety, depression, and kinesiophobia (fear of movement). Kinesiophobia is defined as an excessive and irrational fear of movement due to the belief that it will cause pain or re-injury, and it may further limit mobility and daily functioning.

The aim of this prospective, cross-sectional study is to investigate the prevalence of kinesiophobia among patients with primary knee osteoarthritis and to evaluate its relationship with pain severity and functional capacity. A total of 84 participants aged 40-85 years, diagnosed with knee OA, will be recruited from the Department of Physical Medicine and Rehabilitation, Ankara Training and Research Hospital. Data collection will include demographic and clinical information, quadriceps muscle strength, range of motion, and radiographic staging using the Kellgren-Lawrence scale. Outcome measures include the Tampa Scale for Kinesiophobia (TSK), Visual Analogue Scale (VAS) for pain, and the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) for function.

This study will provide insights into the impact of kinesiophobia on pain and functional outcomes in knee OA and may help guide clinical strategies that address both physical and psychosocial factors in the management of this common condition.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is the most prevalent chronic joint disorder, characterized by progressive cartilage degeneration, abnormal remodeling of the subchondral bone, osteophyte formation, and joint pain that frequently results in disability. The knee joint is particularly vulnerable due to its weight-bearing function and high mechanical stress, making knee OA a leading cause of mobility impairment in older adults. While radiographic evaluation using the Kellgren-Lawrence (K/L) grading system remains the standard method for diagnosing and staging OA, radiographic severity does not always correlate with clinical symptoms such as pain and functional disability. This inconsistency suggests that psychosocial factors may play an important role in shaping the clinical presentation of knee OA.

Kinesiophobia, defined as an excessive and irrational fear of movement due to the anticipation of pain or re-injury, has been reported in various musculoskeletal disorders and post-surgical recovery. High levels of kinesiophobia are associated with worse pain perception, reduced functional capacity, and lower quality of life. In knee OA, the role of kinesiophobia remains controversial, with previous studies reporting inconsistent findings regarding its relationship with pain, functional limitation, and disease progression. Understanding this relationship is crucial, as addressing kinesiophobia may help to optimize rehabilitation outcomes and reduce disability in affected patients.

The present study is a prospective, cross-sectional observational study designed to assess the prevalence of kinesiophobia in patients with primary knee osteoarthritis and to examine its association with pain severity and functional status. A total of 84 patients, aged 40-85 years, with radiographically confirmed knee OA will be recruited from the Department of Physical Medicine and Rehabilitation, Ankara Training and Research Hospital. Patients with prior knee surgery, rheumatological disease, neuromuscular conditions, or systemic inflammatory disorders will be excluded.

Data collection will include demographic variables (age, sex, body mass index, occupation, comorbidities), physical examination findings (range of motion, quadriceps strength), and radiographic staging using the Kellgren-Lawrence scale. Patient-reported outcomes will be assessed using the Visual Analogue Scale (VAS) for pain, the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) for function, and the Tampa Scale for Kinesiophobia (TSK), which has been validated in Turkish populations. Higher scores on these measures indicate greater pain, worse functional limitation, and higher levels of kinesiophobia.

All data will be analyzed using SPSS software. Normality will be assessed using the Kolmogorov-Smirnov test. Depending on data distribution, group comparisons will be made with Student's t test or Mann-Whitney U test, and relationships between kinesiophobia, pain, and function will be explored using correlation and regression analyses. A power analysis determined that a minimum of 84 patients will be required to achieve adequate statistical power at 80%.

By systematically evaluating kinesiophobia alongside clinical and radiographic features of knee OA, this study aims to clarify its role as a psychosocial factor influencing pain and disability. The findings are expected to contribute to improved patient assessment and may support the integration of psychological screening and targeted interventions in the management of knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40-85 years
* Diagnosis of unilateral or bilateral primary knee osteoarthritis
* Duration of knee pain ≥ 3 months
* Radiographic confirmation of tibiofemoral OA (Kellgren-Lawrence grading)

Exclusion Criteria:

* Prior knee surgery
* Deep vein thrombosis
* Neuromuscular disease or neurological disorder
* Mental illness preventing participation
* Active infection or osteomyelitis
* Chronic periarticular infection
* Rheumatologic disease
* Immunodeficiency or systemic inflammatory disease
* Pregnancy

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 40-85 years with radiographically confirmed primary knee osteoarthritis, recruited from the Physical Medicine and Rehabilitation Clinic of Ankara Training and Research Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-30 (Actual)

PRIMARY OUTCOMES:
Kinesiophobia Score (Tampa Scale for Kinesiophobia - TSK) | At baseline, single assessment (Day 1)
  The TSK is a 17-item validated questionnaire assessing fear of movement. Scores range from 17 to 68, with higher scores indicating greater kinesiophobia.

SECONDARY OUTCOMES:
Pain Severity (Visual Analogue Scale - VAS) | At baseline, single assessment (Day 1)
  Pain severity will be measured using a 10 cm-long Visual Analogue Scale (VAS), where 0 = no pain and 10 = worst imaginable pain.
Functional Status (Western Ontario and McMaster Universities Osteoarthritis Index - WOMAC) | At baseline, single assessment (Day 1)
  The WOMAC is a validated 24-item scale assessing pain, stiffness, and physical function. Higher scores indicate greater impairment.
Radiographic Stage (Kellgren-Lawrence Scale) | At baseline, single assessment (Day 1)
  Radiographic severity of knee osteoarthritis will be graded from 0 to 4 according to the Kellgren-Lawrence Scale classification.
Knee Range of Motion (ROM) | At baseline, single assessment (Day 1)
  Measured with a goniometer during physical examination; values reported in degrees.
Quadriceps Muscle Strength | At baseline, single assessment (Day 1)
  Measured using manual muscle testing; results recorded on a 0-5 scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy and Rehabilitation, University of Health Sciences, Ankara Training and Research Hospital, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is observational, involves a single-center hospital population, and collects sensitive clinical and psychosocial information that cannot be adequately de-identified for open sharing. Aggregate results will be reported in publications.

REFERENCES:
- [Background] Canzone A, Roggio F, Patti A, Giustino V, Mannucci C, Di Mauro D, Musumeci G, Bianco A, Trimarchi F. Classification of Physical Activity Programs Based on the Kellgren & Lawrence Scale for Knee Osteoarthritis: A Systematic Review. Musculoskeletal Care. 2024 Dec;22(4):e70019. doi: 10.1002/msc.70019. PMID 39592397
- [Background] Ege F. The relationship between kinesiophobia severity and clinical parameters in patients with mechanical low back pain. J Back Musculoskelet Rehabil. 2024;37(2):285-294. doi: 10.3233/BMR-220365. PMID 37482977
- [Background] Heller GZ, Manuguerra M, Chow R. How to analyze the Visual Analogue Scale: Myths, truths and clinical relevance. Scand J Pain. 2016 Oct;13:67-75. doi: 10.1016/j.sjpain.2016.06.012. Epub 2016 Jul 27. PMID 28850536
- [Background] Peral Perez J, Mortensen SR, Lluch Girbes E, Gronne DT, Thorlund JB, Roos EM, Skou ST. Association between widespread pain and psychosocial factors in people with knee osteoarthritis: a cross-sectional study of patients from primary care in Denmark. Physiother Theory Pract. 2025 Apr;41(4):752-762. doi: 10.1080/09593985.2024.2372381. Epub 2024 Jul 1. PMID 38946473
- [Background] Aydemir B, Huang CH, Foucher KC. Strength and physical activity in osteoarthritis: The mediating role of kinesiophobia. J Orthop Res. 2022 May;40(5):1135-1142. doi: 10.1002/jor.25151. Epub 2021 Aug 6. PMID 34324222
- [Background] Molyneux J, Herrrington L, Riley B, Jones R. A single-arm, non-randomized investigation into the short-term effects and follow-up of a 4-week lower limb exercise programme on kinesiophobia in individuals with knee osteoarthritis. Physiother Res Int. 2020 Jul;25(3):e1831. doi: 10.1002/pri.1831. Epub 2020 Jan 24. PMID 31975503
- [Background] Lisboa FSS, Benevento EM, Kaneko LO, Bertolucci V, Rosini Silva AA, Sardim AC, Ruiz VF, Dos Reis IGM, Porcari AM, Messias LHD. Plasma metabolites associated with biopsychosocial parameters in overweight/obese women with severe knee osteoarthritis. Front Cell Dev Biol. 2024 Sep 4;12:1454084. doi: 10.3389/fcell.2024.1454084. eCollection 2024. PMID 39296935
- [Background] Nedder VJ, Raju AG, Moyal AJ, Calcei JG, Voos JE. Impact of Psychological Factors on Rehabilitation After Anterior Cruciate Ligament Reconstruction: A Systematic Review. Sports Health. 2025 Mar;17(2):291-298. doi: 10.1177/19417381241256930. Epub 2024 Jul 23. PMID 39041333
- [Background] Brown OS, Hu L, Demetriou C, Smith TO, Hing CB. The effects of kinesiophobia on outcome following total knee replacement: a systematic review. Arch Orthop Trauma Surg. 2020 Dec;140(12):2057-2070. doi: 10.1007/s00402-020-03582-5. Epub 2020 Aug 24. PMID 32839826
- [Background] Fischer M, Nonnenmacher L, Sobau C, Zimmerer A. Postoperative hip bracing reduces kinesiophobia in patients undergoing hip arthroscopy: a randomized-controlled trial. Arch Orthop Trauma Surg. 2024 Jul;144(7):3205-3210. doi: 10.1007/s00402-024-05437-9. Epub 2024 Jul 9. PMID 38980377
- [Background] Han S, Oh M, Lee H, Hopkins JT. The effects of kinesiophobia on postural control with chronic ankle instability. Gait Posture. 2024 Jan;107:269-274. doi: 10.1016/j.gaitpost.2023.10.014. Epub 2023 Oct 18. PMID 37914561
- [Background] Reddy RS, Alshahrani MS, Tedla JS, Dixit S, Gular K, Kakaraparthi VN. Exploring the Interplay Between Kinesiophobia, Lumbar Joint Position Sense, Postural Stability, and Pain in Individuals With Chronic Low Back Pain: A Cross-Sectional Analysis. J Manipulative Physiol Ther. 2023 Jun-Dec;46(5-9):294-304. doi: 10.1016/j.jmpt.2024.09.004. Epub 2024 Oct 16. PMID 39425703
- [Background] Asiri F, Reddy RS, Tedla JS, ALMohiza MA, Alshahrani MS, Govindappa SC, Sangadala DR. Kinesiophobia and its correlations with pain, proprioception, and functional performance among individuals with chronic neck pain. PLoS One. 2021 Jul 8;16(7):e0254262. doi: 10.1371/journal.pone.0254262. eCollection 2021. PMID 34237105
- [Background] Luque-Suarez A, Martinez-Calderon J, Falla D. Role of kinesiophobia on pain, disability and quality of life in people suffering from chronic musculoskeletal pain: a systematic review. Br J Sports Med. 2019 May;53(9):554-559. doi: 10.1136/bjsports-2017-098673. Epub 2018 Apr 17. PMID 29666064
- [Background] Lozano-Meca J, Gacto-Sanchez M, Montilla-Herrador J. Association of kinesiophobia with pain, disability and functional limitation in adults with knee osteoarthritis: A systematic review and meta-analysis. Geriatr Nurs. 2024 Nov-Dec;60:481-490. doi: 10.1016/j.gerinurse.2024.10.013. Epub 2024 Oct 18. PMID 39426272
- [Background] Jang S, Lee K, Ju JH. Recent Updates of Diagnosis, Pathophysiology, and Treatment on Osteoarthritis of the Knee. Int J Mol Sci. 2021 Mar 5;22(5):2619. doi: 10.3390/ijms22052619. PMID 33807695
- [Background] Wu Q, Xu Z, Ma X, Li J, Du J, Ji J, Ling X, Kan J, Zhao M. Association of low muscle mass index and sarcopenic obesity with knee osteoarthritis: a systematic review and meta-analysis. J Int Soc Sports Nutr. 2024 Dec;21(1):2352393. doi: 10.1080/15502783.2024.2352393. Epub 2024 May 22. PMID 38775452